CLINICAL TRIAL: NCT05394077
Title: Effect of Active Release Technique and Abdominal Drawing-Maneuver on Pain and Quality of Life in Patients With Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall17/518
Record Dates: First submitted 2022-05-09; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Release Technique (Experimental): Using Active Release Technique
  Interventions: Diagnostic Test: Active Release Technique
- Abdominal Drawing-Maneuver (Experimental): Using Abdominal Drawing-Maneuver Technique
  Interventions: Diagnostic Test: Abdominal Drawing-Maneuver

INTERVENTIONS:
Diagnostic Test: Active Release Technique — Using Active Release Technique
  Arms: Active Release Technique
Diagnostic Test: Abdominal Drawing-Maneuver — Using Abdominal Drawing-Maneuver Technique
  Arms: Abdominal Drawing-Maneuver

SUMMARY:
To determine the effect of active release technique and abdominal drawing in maneuver on pain and quality of life in patients of chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient with hamstring tightness[9]
* Subjects with pain between 4 and 7cm on visual analogue scale[18].
* Subjects having 20-40 age group are included in this study[11]
* Patients having pain for more than 3 month of mild-moderate intensity[9]

Exclusion Criteria:

* Patients with any spine injury[11]
* Lumber intervertebral disc fracture[11]
* Patients having any surgical history of spine[11]
* Spinal stenosis[11]

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Abdominal Drawing-Maneuver on Pain and Quality of Life in Patients With Chronic Low Back Pain | 6 Months
  11 participents with The Hot pack initially for 10 minutes then this group will receive abdominal drawing-in maneuver technique for 2 times in week of 10 session. SF-36 Questionnaire.

SECONDARY OUTCOMES:
Active Release Technique in Patients With Chronic Low Back Pain | 6 Months
  12 participents with The Hot pack initially for 10 minthen this group will receive active release technique 2 times in week of 10 session while other group will receive abdominal drawing-in maneuver technique for 2 times in week of 10 session. Visual analogue scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Ibrahim PT Clinic Lahore Zohaib Physiotherapy Clinic, Farooq Abad, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No